CLINICAL TRIAL: NCT06908603
Title: Use of Artificial Intelligence in Oral Radiology: A Multicenter Cross-Sectional Study in Egypt
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora Saif Taha, Associate Professor, Oral & Maxillofacial Radiology, Faculty of Dentistry, Cairo University, Cairo University
Other Study IDs: EMRALab_001
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Knowledge of AI Applications in Dental Imaging
Keywords: AI; AI knowledge; AI perception; dentistry; oral radiology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Survey using a questionnaire. — The online, self-administered, 16-item questionnaire included several question styles (yes/no questions, closed-ended, multiple choice questions, and statements with Likert scale responses). The questionnaire was adapted from several published AI surveys . Questions were designed to assess three primary areas: AI knowledge, perceptions of AI integration into practice and challenges in implementing AI in the OR practice in Egypt.

SUMMARY:
The survey aims to assess knowledge and perceptions of AI applications in dental imaging among Egyptian dentists. It also aims to identify the needs and challenges of implementing this transformative technology into education, training, and clinical practice.

DETAILED DESCRIPTION:
Artificial Intelligence (AI) is advancing rapidly in the field of dentistry, particularly in diagnostic imaging. These AI-based tools are aiding dentists by making it easier to detect important structures and identify health issues with greater accuracy. Dentists around the world, including those in Egypt, are gradually integrating AI into oral radiology. However, the successful use of AI depends heavily on the dentists being aware and prepared to use it effectively. The Egyptian government is very keen on incorporating AI into healthcare and has developed programs like the National Artificial Intelligence Strategy to promote its use. Despite these efforts, research on Egyptian dentists' comprehension and views about AI in oral radiology is still limited. The study seeks to evaluate Egyptian dentists' knowledge about AI and to uncover the primary obstacles that prevent them from utilizing AI effectively in clinical settings.

A cross-sectional survey was conducted online among Egyptian dentists. The questionnaire aimed to assess their knowledge, attitudes, and perceived challenges related to AI in oral radiology. Dentists were recruited through academic institutions, professional organizations, and social media platforms. To identify factors influencing respondents' knowledge about AI, a logistic regression analysis was applied.

ELIGIBILITY:
Inclusion Criteria:

* graduated dentists with a bachelor's or higher degree from Egyptian universities who practiced in Egypt.

Exclusion Criteria:

* Undergraduate students and dentists who obtained their undergraduate qualification abroad or practiced outside Egypt were excluded.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Faculty members and postgraduate dental students at the Faculty of Dentistry, Cairo University, as well as members of the Egyptian Maxillofacial Radiology Alliance from various academic dental institutions across Egypt, including Alexandria University, Ain Shams University, Al-Azhar University, Beni-Suef University, Misr International University, Future University in Egypt, Misr University for Science and Technology, and British University in Egypt. Additionally, social media platforms were utilized to engage members of other Egyptian dental societies.
Sampling Method: Non-Probability Sample
Enrollment: 1326 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Assessment of the reported level of knowledge of AI applications in dental imaging using a standardized questionnaire | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eschert T, Schwendicke F, Krois J, Bohner L, Vinayahalingam S, Hanisch M. A Survey on the Use of Artificial Intelligence by Clinicians in Dentistry and Oral and Maxillofacial Surgery. Medicina (Kaunas). 2022 Aug 5;58(8):1059. doi: 10.3390/medicina58081059. PMID 36013526